CLINICAL TRIAL: NCT03345342
Title: A Double-blind, Randomized, Active-controlled, Parallel-group Study of Paliperidone Palmitate 6-Month Formulation
Brief Title: A Study of Paliperidone Palmitate 6-Month Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108390; R092670PSY3015 (Other: Janssen Research & Development, LLC); 2017-001941-28 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- PP1M: Transition Phase (Experimental): Participants who previously have not achieved stability with moderate to higher doses of Paliperidone palmitate 1-month (PP1M) or Paliperidone palmitate 3-month (PP3M) will enter into a transition period of up to 4 months. During transition period participants will receive 1 to 5 injections of PP1M 50 to 100 milligrams equivalent (mg eq.). The participants who achieved stability (stability is defined as at least 3 months of injections with the last 2 doses being the same strength) with PP1M 100 mg eq. will precede from transition phase to maintenance phase.
  Interventions: Drug: PP1M
- PP1M/PP3M: Maintenance Phase (Experimental): All the participants will receive only 1 dose of PP1M 100 or 150 mg eq. or PP3M 350 or 525 mg eq. The participants will precede from maintenance phase to double-blind phase.
  Interventions: Drug: PP3M 350 mg eq.; Drug: PP3M 525 mg eq.; Drug: PP1M
- PP6M or Placebo: Double-Blind Phase (Experimental): Participants will receive intramuscular injection of PP6M in left gluteal muscle on Day 1 and right gluteal muscle on Day 183 with alternating placebo in right gluteal muscle on Day 92 and left gluteal muscle on Day 274.
  Interventions: Drug: PP6M; Other: Placebo
- PP3M: Double-Blind Phase (Experimental): Participants will receive intramuscular injections of PP3M at dose of 350 mg eq. or 525 mg eq. in left gluteal muscle on Day 1 and 274 and right gluteal muscle on Day 92 and 183.
  Interventions: Drug: PP3M 350 mg eq.; Drug: PP3M 525 mg eq.

INTERVENTIONS:
Drug: PP6M — Participants will receive intramuscular injection of PP6M.
  Other Names: R092670
  Arms: PP6M or Placebo: Double-Blind Phase
Drug: PP3M 350 mg eq. — Participants will receive intramuscular injection of PP3M 350 mg eq.
  Other Names: R092670
  Arms: PP1M/PP3M: Maintenance Phase; PP3M: Double-Blind Phase
Drug: PP3M 525 mg eq. — Participants will receive intramuscular injection of PP3M 525 mg eq.
  Other Names: R092670
  Arms: PP1M/PP3M: Maintenance Phase; PP3M: Double-Blind Phase
Drug: PP1M — Participants will receive intramuscular injection of PP1M 50 to 150 mg eq.
  Other Names: R092670
  Arms: PP1M/PP3M: Maintenance Phase; PP1M: Transition Phase
Other: Placebo — Participants will receive matching placebo.
  Arms: PP6M or Placebo: Double-Blind Phase

SUMMARY:
The purpose of this study is to demonstrate that injection cycles consisting of a single administration of paliperidone palmitate 6-month (PP6M) are not less effective than 2 sequentially administered injections of paliperidone palmitate 3-month PP3M) (350 or 525 mg eq.) for the prevention of relapse in participants with schizophrenia previously stabilized on corresponding doses of paliperidone palmitate 1-month (PP1M) (100 or 150 mg eq.) or PP3M (350 or 525 mg eq.).

DETAILED DESCRIPTION:
The primary hypothesis of this study is that the efficacy of PP6M is non-inferior to PP3M for preventing relapse in participants with schizophrenia who were previously stabilized on corresponding doses of PP1M or PP3M. The study consists of mainly 3 phases: a screening phase (up to 28 days), a maintenance phase (of 1 or 3 months), and a double-blind phase (of 12 months [neither the researchers nor the participants know what treatment the participant is receiving]). Additional/conditional phases include a transition phase (before maintenance phase). Study evaluations include efficacy, pharmacokinetics, pharmacodynamics, and safety. The study duration will vary from approximately 13 months to 19 months.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) for at least 6 months before screening
* Must be receiving treatment with paliperidone palmitate (as either the paliperidone palmitate 1-month (PP1M) or paliperidone palmitate 3-month (PP3M) formulation), or injectable risperidone, or any oral antipsychotic
* Must be able, in the opinion of the investigator, to discontinue any antipsychotic medication other than PP1M) or PP3M during the Screening Phase
* Must have a full Positive and Negative Syndrome Scale (PANSS) score of less than (<) 70 points at screening
* Must have a body mass index (BMI) between 17 and 40 kilogram (kg)/meter (m)^2 (inclusive) and must have a body weight of at least 47 kg at screening
* Must be willing to receive gluteal injections of medication during the Double-blind Phase

Exclusion Criteria

* Must not be receiving any form of involuntary treatment, such as involuntary psychiatric hospitalization, parole-mandated treatment, or court-mandated treatment
* Must not have attempted suicide within 12 months before screening and must not be at imminent risk of suicide or violent behavior, as clinically assessed by the investigator at the time of screening
* Must not have a DSM-5 diagnosis of moderate or severe substance use disorder (except for nicotine and caffeine) within 6 months of screening; however, acute or intermittent substance use prior to screening is not exclusionary, depending upon the clinical judgment of the investigator
* Must not have a history of neuroleptic malignant syndrome or tardive dyskinesia
* Must not have a history of intolerability or severe reactions to moderate or higher doses of antipsychotic medications and must not have any other factors that would, in the judgment of the investigator, indicate that treatment with moderate or higher doses of paliperidone palmitate would be intolerable or unsafe

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (138):
- United States (25):
  - Woodland Research Northwest, Rogers, Arkansas
  - California Pharmaceutical Research Institute, Inc., Anaheim, California
  - ATP Clinical Research, Costa Mesa, California
  - Collaborative NeuroScience Network, Garden Grove, California
  - Synergy East, Lemon Grove, California
  - Pacific Research Partners, Oakland, California
  - SF-Care, Inc, San Rafael, California
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Clintex Research Group, Miami, Florida
  - Florida Research Center Inc., Miami, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Alexian Behavioral Health Hospital, Hoffman Estates, Illinois
  - Ascension via Christi Research, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cherry Street Services, Inc., Grand Rapids, Michigan
  - St. Louis Clinical Trials, St Louis, Missouri
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Clinical Trials of America Inc, Hickory, North Carolina
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Future Search Trials of Dallas, Dallas, Texas
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
- Argentina (6):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - CEN, Córdoba
  - Sanatorio Prof. Leon S. Morra, Córdoba
  - Instituto de Neurociencias San Agustin, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
- Australia (2):
  - The Lyell McEwin Hospital, Elizabeth Vale
  - Neuro Trials Victoria, Noble Park
- Brazil (7):
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Instituto Bairral de Psiquiatria, Itapira
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Bulgaria (6):
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - State Psychiatric Hospital Pazardzhik, Pazardzhik
  - UMHAT 'Sveti Georgi'-Plovdiv, Plovdiv
  - State Psychiatric HospitalDr.Georgi Kissiov, Radnevo
  - Centre for Mental Health Prof.N.Shipkovenski EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
- Czechia (6):
  - Psychiatricka ambulance, MUDr. Marta Holanova, Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Kralove-Vekose
  - A Shine S R O, Pilsen
  - Pragtis S R O, Prague
  - Institut Neuropsychiatricke pece, Prague
  - Psychiatricka ambulance MUDr. Simona Papezova, Prague
- France (5):
  - C.H.S. Charles Perrens, Bordeaux
  - CHRU La Colombière, Montpellier
  - CHU Caremeau, Nîmes
  - Hopital Sainte Anne, Paris
  - Hopital Sainte Musse, Toulon
- Hong Kong (2):
  - Kwai Chung Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (4):
  - Józsefvarosi Szent Kozma Egészségügyi Központ, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bács-Kiskun Megyei Kórház a Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, Kalocsa
  - CRU Hungary Kft., Miskolc
- India (8):
  - Ratandeep Multispeciality Hospital, Ahmedabad
  - Sri Ramachandra Medical Centre, Chennai
  - Asha hospital, Hyderabad
  - Ahana Hospitals, Madurai
  - Vinaya Hospital and Research Center, Mangalore
  - Kasturba Medical College Hospital, Manipal
  - Jehangir Clinical Development Center Pvt Ltd, Pune
  - Deva Institute of Health Care and Research Pvt Ltd, Varanasi
- Italy (4):
  - Clinica Psichiatrica - Università di Cagliari, Cagliari
  - Dipartimento di Salute Mentale, Lecce
  - Seconda Universita degli Studi di Napoli - Azienda Ospedaliera Universitaria, Napoli
  - Universita degli Studi di Roma 'La Sapienza' - Azienda Ospedaliera Sant Andrea, Roma
- Malaysia (4):
  - Hospital Bahagia Ulu Kinta, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Mexico (5):
  - Gabipros SC, Mexico City
  - Instituto Neuropsique, Monterrey
  - Centro de Estudios Clinicos y Especialidades Medicas S C, Monterrey
  - Infosame/Research, Monterrey
  - Centro de Atencion e Investigacion Cardiovascular del Potosi S C, San Luis Potosí City
- Poland (10):
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Wlokiennicza MED Specjalistyczna Praktyka Lekarska dr n.med. Tomasz Markowski, Bialystok
  - Zespol Opieki Zdrowotnej w Chelmnie, Chełmno
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Szpital Specjalistyczny im H Klimontowicza Oddzial Psychiatryczny, Gorlice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Centrum Medyczne Luxmed Sp z o o, Lublin
  - Poradnia Zdrowia Psychicznego 'Syntonia' w Pruszczu Gdanskim, Pruszcz Gdański
  - Mazowieckie Specjalistyczne Centrum Zdrowia im. Prof. Jana Mazurkiewicza w Pruszkowie, Pruszków
  - Wojewodzki Szpital Zespolony im L Rydygiera w Toruniu, Torun
- Russia (12):
  - Clinical Psychiatric Hospital #3 Named After V.A. Gilyarovsky, Moscow
  - Psychiatric Clinical hospital 1 named after N.A. Alekseev, Moscow
  - Nizny Novgorod clinical psychiatric hospital 1, Nizny Novgorod
  - Psychoneurological Dispensary of Frunzensky District, Saint Petersburg
  - Psychoneurological dispensary 10, Saint Petersburg
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - Psychoneurological dispensary 1, Saint Petersburg
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Saratov Regional Psychiatric hospital named after St. Sofia, Saratov
  - Psychoneurological Dispensary #4, St.Peterburg
  - Research Institute of Mental Health, Tomsk
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg
- South Africa (3):
  - Flexivest 14 Research, Cape Town
  - Gert Bosch Pretoria South Africa, Pretoria
  - Juan Schrönen - Western Cape South Africa, Welgemoed
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Chonbuk National Univ Hospital, Jeonju
  - Seoul National University Hospital, Seoul
- Spain (7):
  - Hosp Univ Vall D Hebron, Barcelona
  - Inst. Internac. Neurociencias Aplicadas, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Centro Salud Mental La Corredoria, Oviedo
  - Hosp. El Bierzo, Ponferrada
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Prov. de Zamora, Zamora
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (5):
  - Abdurrah Yurtarslan Training and Research Hospital, Ankara
  - Ankara Numune Research and Training Hospital, Ankara
  - Erenkoy Mental Health Hospital, Istanbul
  - Selcuk University, Medical School, Department of Psychiatry, Konya
  - Sakarya University Medical Faculty Psychiatry Department, Sakarya
- Ukraine (9):
  - MNCE of Kyiv RC Regional Psychiatric and Narcological Medical Association, Hlevakha
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - CNPE'Kherson Regional Institution of Mental Care'of Kherson Regional Council, Kherson
  - Kyiv Territorial Medical Incorporation 'Psychiatry', Kyiv
  - Municipal Institution 'Lviv Regional Clinical Psycho-Neurological Dispensary', Lviv
  - CNCE of the Lviv Regional Council 'Lviv Regional Clinical Psychiatric Hospital', Lviv
  - CNCE Odesa regional psychiatric hospital #2 Odesa regional council, Oleksandrivka
  - CNCE 'Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council', Smila
  - CNCE 'Vinnytsya RC Psychoneurological Hospital n.a. O.I. Yushchenko Vinnytsya RC', Vinnytsia

REFERENCES:
- [Derived] Richarz U, Han J, Bai YM, Yu-Hai Chen E, Chung YC, Jhanwar VG, Kim SW, Sulaiman AH, Knight K, Gopal S. Efficacy and safety of paliperidone palmitate 6-monthly long-acting injectable in reduction of relapses in patients with schizophrenia: An Asian subgroup analysis of phase 3, randomized study. Medicine (Baltimore). 2023 Aug 25;102(34):e34623. doi: 10.1097/MD.0000000000034623. PMID 37653768
- [Derived] Najarian D, Turkoz I, Knight RK, Galderisi S, Lamaison HF, Zalitacz P, Aravind S, Richarz U. Long-Term Efficacy and Safety of Paliperidone 6-Month Formulation: An Open-Label 2-Year Extension of a 1-Year Double-Blind Study in Adult Participants With Schizophrenia. Int J Neuropsychopharmacol. 2023 Aug 29;26(8):537-544. doi: 10.1093/ijnp/pyad028. PMID 37480362
- [Derived] Najarian D, Sanga P, Wang S, Lim P, Singh A, Robertson MJ, Cohen K, Schotte A, Milz R, Venkatasubramanian R, T'Jollyn H, Walling DP, Galderisi S, Gopal S. A Randomized, Double-Blind, Multicenter, Noninferiority Study Comparing Paliperidone Palmitate 6-Month Versus the 3-Month Long-Acting Injectable in Patients With Schizophrenia. Int J Neuropsychopharmacol. 2022 Mar 17;25(3):238-251. doi: 10.1093/ijnp/pyab071. PMID 34791283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 841 participants were enrolled, out of which 838 participants received treatment. 2 participants were enrolled but did not receive treatment and 1 participant withdrew from the Open-label Phase and as permitted per the protocol, re-entered the study (under a different participant identifier) and was counted twice in the total. Per the rules specified in statistical analysis plan, only data collected during the second study participation was included in data summary for this participant.
Groups:
- Open-Label (OL) PP1M/PP3M: Participants previously treated with oral antipsychotics, or injectable risperidone, or a moderate or higher dose of paliperidone palmitate 1-month (PP1M) with previous initiation but without previous stabilization (where stabilization was defined as at least 3 months of injections with the last 2 doses being the same strength) received 1 to 5 intramuscular (IM) injections of PP1M 50 to 150 milligrams equivalent (mg eq.). Participants received single dose of IM injection of PP1M as 100 or 150 mg eq. or PP3M as 350 or 525 mg eq during the OL-maintenance phase.
- Double-blind PP3M: Participants received 4 doses of PP3M (350 or 525 mg eq. IM injection for up to 12 months (1 dose every 3 month) during DB phase.
- Double-blind PP6M: Participants received 2 doses of PP6M (700 or 1000 mg eq. IM injection for 12 months (1 dose every 6 months), during the DB Phase. To maintain blinding, participants received IM injections of matching placebo at the 3-month time points between their 6-month doses of PP6M drug.
- Follow-up (FU) Phase PP3M: Participants who have received at least 1 dose of PP3M (350 or 525 mg eq.) IM injection during double-blind phase but then have relapsed or have met other relevant conditions for withdrawal or discontinuation can participate in the follow-up phase PP3M (350 or 525 mg eq.) IM injection for up to 12 months for evaluating efficacy and safety.
- Follow-up Phase PP6M: Participants received PP6M (700 or 1000 mg eq.) IM injection for up to 12 months for evaluating efficacy and safety.
Period: Open-Label Phase
Arm/Group | Open-Label (OL) PP1M/PP3M | Double-blind PP3M | Double-blind PP6M | Follow-up (FU) Phase PP3M | Follow-up Phase PP6M
Started | 838 | 0 | 0 | 0 | 0
Completed | 702 | 0 | 0 | 0 | 0
Not Completed | 136 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 30 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Initiated Prohibited Medication | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0 | 0
Not completed — Non-Compliance with Study Drug | 4 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 57 | 0 | 0 | 0 | 0
Not completed — Other | 15 | 0 | 0 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Open-Label (OL) PP1M/PP3M | Double-blind PP3M | Double-blind PP6M | Follow-up (FU) Phase PP3M | Follow-up Phase PP6M
Started | 0 | 224 (Participants from the OL phase have continued in the DB phase.) | 478 (Participants from the OL phase have continued in the DB phase.) | 0 | 0
Completed | 0 | 202 | 416 | 0 | 0
Not Completed | 0 | 22 | 62 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 6 | 0 | 0
Not completed — Death | 0 | 2 | 1 | 0 | 0
Not completed — Initiated Prohibited Medication | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 7 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 16 | 38 | 0 | 0
Not completed — Other | 0 | 1 | 3 | 0 | 0
Period: Follow-Up Phase
Arm/Group | Open-Label (OL) PP1M/PP3M | Double-blind PP3M | Double-blind PP6M | Follow-up (FU) Phase PP3M | Follow-up Phase PP6M
Started | 0 | 0 | 0 | 42 (Participants from the DB phase have continued in the FU phase.) | 109 (Participants from the DB phase have continued in the FU phase.)
Completed | 0 | 0 | 0 | 34 | 78
Not Completed | 0 | 0 | 0 | 8 | 31
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 15
Not completed — Other | 0 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label (OL) PP1M/PP3M
Number analyzed (Participants) | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285
  Male | 553
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118
  Not Hispanic or Latino | 710
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 111
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 106
  White | 606
  More than one race | 5
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 55
  AUSTRALIA | 4
  BRAZIL | 90
  BULGARIA | 46
  CZECH REPUBLIC | 45
  FRANCE | 7
  HONG KONG | 4
  HUNGARY | 20
  INDIA | 42
  ITALY | 8
  KOREA, REPUBLIC OF | 4
  MALAYSIA | 22
  MEXICO | 23
  POLAND | 68
  RUSSIAN FEDERATION | 139
  SPAIN | 29
  TAIWAN | 31
  TURKEY | 26
  UKRAINE | 50
  UNITED STATES | 125

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse During the Double-Blind (DB) Phase
Description: Time to relapse is time between participant randomization in DB Phase and first documentation of relapse event by end of Month 12 of DB phase. Relapse is defined as: a) Psychiatric hospitalization; b) Positive and Negative Syndrome Scale (PANSS) total score: Increase of 25 percentage (%), 10 point increase in PANSS for 2 analysis separated by 3-7 days if score was greater than (>) 40, less than or equal to (<=)40; c) Participants inflicted knowing self-injury/shown violent behavior leading to suicide, clinically significant injury to him/herself or other person/property; d) Participants had suicidal/homicidal ideation/violent behavior that was clinically significant as per investigator; e) PANSS items P1- delusions, P2- conceptual disorganization, P3-hallucinatory behavior, P6- suspiciousness/ persecution, P7-hostility, G8-uncooperativeness: score: greater than or equal to (>=)5, >=6 for 2 analysis separated by 3-7 days on any items if maximum score for PANSS: <=3 or 4, respectively.
Time Frame: Up to 12 months of DB Phase
Population: DB Intent-to-Treat (ITT) analysis set included participants who were randomly assigned to paliperidone palmitate 6-month (PP6M) /paliperidone palmitate 3-month (PP3M) during DB Phase, received at least 1 dose of PP6M/PP3M.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- DB PP3M: Participants received 4 doses of PP3M (350 or 525 milligrams equivalent [mg eq.]) intramuscular (IM) injection for up to 12 months (1 dose every 3 month) during DB phase.
- DB PP6M: Participants received 2 doses of PP6M (700 or 1000 mg eq.) IM injection for 12 months (1 dose every 6 months), during the DB Phase. To maintain blinding, participants received IM injections of matching placebo at the 3-month time points between their 6-month doses of PP6M drug.
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 224 | 478
Days | NA [NA to NA] — NA indicates that the median, lower and upper limit of confidence interval (CI) was not estimable due to insufficient number of events to determine this value. | NA [NA to NA] — NA indicates that the median, lower and upper limit of confidence interval (CI) was not estimable due to insufficient number of events to determine this value.

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The neuropsychiatric symptoms of schizophrenia were assessed using the 30-item PANSS scale, which provides a total score (sum of the scores for all 30 items) and scores for 3 subscales: the 7-item positive-symptom (P) subscale, the 7-item negative-symptom (N) subscale, and the 16-item general-psychopathology symptom (G) subscale. Each item is rated on a scale from 1 (absent) to 7 (extreme). The PANSS total score ranges from 30 (absent disease)-210 (more severe neuropsychiatric symptoms of schizophrenia).
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: DB ITT analysis set included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M. Here 'N' (number of participants analyzed), signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DB PP3M: Participants received 4 doses of PP3M (350 or 525 mg eq.) IM injection for up to 12 months (1 dose every 3 month) during DB phase.
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 220 | 473
units on a scale | -1.6 (7.40) | -1.8 (8.92)

3. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity (CGI-S) Score
Description: CGI-S is defined as clinician-rated scale that assesses the severity of mental illness on a scale of 0 to 7. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating according to:1: normal, not at all ill; 2: borderline mentally ill; 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; 7: among the most extremely ill patients. A higher score implies a more severe condition.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: DB ITT analysis set included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 221 | 475
units on a scale | 0.0 (0.63) | 0.0 (0.70)

4. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Scale Total Score
Description: The Personal and Social Performance (PSP) scale assesses degree of a participant's dysfunction within 4 domains of behavior: 1) socially useful activities, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior. Each domain was assessed on a 6-point scale, from 1 (absent) to 6 (very severe) (1 = absent, 2 = mild, 3 = manifest, 4 = marked, 5 = severe, and 6 = very severe). PSP total score was calculated as sum of all the domain scores and ranges from 1 to 100. Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision. Higher score indicates better performance.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 220 | 473
units on a scale | 1.1 (8.11) | 1.0 (7.12)

5. Secondary Outcome: Percentage of Participants With Symptomatic Remission Based on PANSS Score During DB Phase
Description: Symptomatic remission was defined as achieving intensity level of mild or moderate on PANSS scale by all 8 items as the determinants for symptomatic remission: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, lack of spontaneity. The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent), 2 (minimal), 3 (mild), 4 (moderate), 5 (moderately severe), 6 (severe) and 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.
Time Frame: Up to 12 months of DB Phase
Population: DB ITT included all participants who were randomly assigned to treatment group of either PP6M or PP3M, received at least 1 dose of PP6M/PP3M.
Measure: Number; unit: Percentage of participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 224 | 478
Percentage of participants | 70.1 | 66.3

6. Secondary Outcome: Change From Baseline in the Satisfaction With Participants in Social Roles (SPSR) Score
Description: The SPSR Short Form 8a is a participant-reported outcome used to assess the satisfaction with participation in social roles. The participants were asked to rate 8 items on 5-point Likert scale, with scores ranging from 8 to 40, where higher scores represents higher satisfaction.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 70 | 154
units on a scale | 0.9 (7.15) | 0.6 (6.58)

7. Secondary Outcome: Change From Baseline in the Treatment Satisfaction Questionnaire for Medication (TSQM-9) Total Score
Description: TSQM-9 consists of 9 questions to assess patients' satisfaction with medication using a range of responses from 1 (extremely dissatisfied) to (7 extremely satisfied). This patient reported outcome provides scores on three parts: effectiveness, convenience, and global satisfaction. The sum of the 9-questions were calculated and used for analysis. The total score ranges from 0 to 63, with higher scores indicating better treatment satisfaction.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 121 | 279
units on a scale
  Effectiveness | 6.0 (21.18) | 3.6 (19.49)
  Convenience | 3.4 (17.76) | 1.1 (15.30)
  Overall satisfaction | 2.5 (19.29) | 0.5 (20.02)

8. Secondary Outcome: Change From Baseline in the Simpson-Angus Rating Scale (SAS) Total Score
Description: The SAS rates 10 items for general extrapyramidal symptoms (EPS) on a 5-point scale from 0 (normal) to 4 (extreme), including gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head rotation, Glabellar tap, tremor, and salivation. The SAS total score is the average score (total sum of item scores divided by the number of items) and ranges between 0 and 4. Negative change in score indicates improvement. Higher scores denote more severe condition of EPS.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 220 | 477
units on a scale | 0.00 [-0.6 to 2.1] | 0.00 [-0.6 to 1.5]

9. Secondary Outcome: Number of Participants With Symptoms of Akathisia Assessed Using Barnes Akathisia Rating Scale (BARS) Score
Description: BARS is used to rate observable, restless movements of drug induced akathisia and subjective awareness of restlessness and any distress associated with the akathisia. BARS consists of the following 4 items: objective assessment of akathisia symptoms, subjective assessment of the participants's awareness of inner restlessness, distress restlessness, and global clinical assessment of akathisia. First three items are rated on a 4-point scale ranging from 0 (no abnormal movements or absence of inner restlessness or no distress) to 3 (severe akathisia or awareness of intense compulsion to move most of the time or severe distress). The last item, the global clinical assessment of akathisia, is rated on a 6-point scale, ranging from 0 (no evidence of akathisia) to 5 (severe akathisia).
Time Frame: Up to 12 Months of DB Phase
Population: DB ITT analysis set included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M.
Measure: Count of Participants; unit: Participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 224 | 478
Participants
  Global Clinical Assessment | 185 | 380
  Objective | 185 | 380
  Subjective (Awareness) | 185 | 380
  Subjective (Distress) | 185 | 380

10. Secondary Outcome: Change From Baseline in the Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: AIMS is a 14-item scale. Items 1 to 8 are rated on a 5-point scale ranging from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Item 9 assesses the participant's incapacitation due to abnormal movements, and item 10 assesses the participant's awareness of the abnormal movements and associated distress. Items 9 and 10 are rated on 5-point scales ranging from 0 (none or no awareness) to 4 (severe or aware, severe distress). Items 11 to 14 are yes/no questions regarding the global judgement and dental status of the participant. The total score is the sum of the scores for the 14 items and the possible total score ranges from 0 to 44. A higher total score is indicative of more severe dyskinetic movements.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Groups:
- Double-blind (DB) PP3M: Participants received 4 doses of PP3M (350 or 525 mg eq.) IM injection for up to 12 months (1 dose every 3 month) during DB phase.
- Double-blind (DB) PP6M: Participants received 2 doses of PP6M (700 or 1000 mg eq.) IM injection for 12 months (1 dose every 6 months), during the DB Phase. To maintain blinding, participants received IM injections of matching placebo at the 3-month time points between their 6-month doses of PP6M drug.
Arm/Group | Double-blind (DB) PP3M | Double-blind (DB) PP6M
Number analyzed (Participants) | 221 | 477
units on a scale | 0.0 [-3 to 2] | 0.0 [-7 to 14]

11. Secondary Outcome: Number of Participants Based on Columbia Suicide Severity Rating Scale (C-SSRS) Total Score
Description: The C-SSRS is a questionnaire used for suicide risk assessment. Affirmative or negative responses are provided to items 1 to 5 for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods [not plan] without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and items 6 to 10 for suicide behavior (6. Preparatory acts or behavior, 7. Aborted attempt, 8. Interrupted attempt, 9. Actual attempt, 10. Completed suicide). Total score ranges from 1 to 10. Higher scores indicate more severe suicidal ideation.
Time Frame: Baseline and endpoint (12 Months of DB Phase)
Population: DB ITT analysis set included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M. Here 'n' (number analyzed) included all evaluable participants who were analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 224 | 478
Participants
  Baseline (0= No event) | 221 | 477
  Baseline (1= Wish to be dead) | 3 | 0
  Baseline (2= Non-specific suicidal thought) | 0 | 1
  Baseline (3= Suicidal ideation-no intent) | 0 | 0
  Baseline (4= Ideation with intent, no plan) | 0 | 0
  Baseline (5= Ideation with plan/intent) | 0 | 0
  Baseline (6= Preparatory acts/behavior) | 0 | 0
  Baseline (7= Aborted attempt) | 0 | 0
  Baseline (8= Interrupted attempt) | 0 | 0
  Baseline (9= Actual attempt) | 0 | 0
  Baseline (10= Suicide) | 0 | 0
  End Point (0= No event): number analyzed (Participants) | 221 | 476
  End Point (0= No event) | 218 | 471
  End Point (1= Wish to be dead): number analyzed (Participants) | 221 | 476
  End Point (1= Wish to be dead) | 1 | 1
  End Point (2= Non-specific suicidal thought): number analyzed (Participants) | 221 | 476
  End Point (2= Non-specific suicidal thought) | 0 | 0
  End Point (3= Suicidal ideation-no intent): number analyzed (Participants) | 221 | 476
  End Point (3= Suicidal ideation-no intent) | 0 | 1
  End Point (4= Ideation with intent, no plan): number analyzed (Participants) | 221 | 476
  End Point (4= Ideation with intent, no plan) | 1 | 0
  End Point (5= Ideation with plan/intent): number analyzed (Participants) | 221 | 476
  End Point (5= Ideation with plan/intent) | 1 | 2
  End Point (6= Preparatory acts/behavior): number analyzed (Participants) | 221 | 476
  End Point (6= Preparatory acts/behavior) | 0 | 0
  End Point (7= Aborted attempt): number analyzed (Participants) | 221 | 476
  End Point (7= Aborted attempt) | 0 | 0
  End Point (8= Interrupted attempt): number analyzed (Participants) | 221 | 476
  End Point (8= Interrupted attempt) | 0 | 0
  End Point (9= Actual attempt): number analyzed (Participants) | 221 | 476
  End Point (9= Actual attempt) | 0 | 1
  End Point (10= Suicide): number analyzed (Participants) | 221 | 476
  End Point (10= Suicide) | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal Electrocardiogram (ECG) Values During DB Phase
Description: Number of participants with treatment-emergent abnormal ECG values were reported. It includes heart rate (abnormally low refers to less than or equal to [<=] 50 beats per minute (bpm) , abnormally high refers greater than or equal to [>=] 100 bpm), pulse rate (PR) interval (abnormally high refers to >= 210 milliseconds [msec]), QRS interval (abnormally Low refers to <= 50, abnormally high refers to >= 120 msec) and QT interval (abnormally low refers to <= 200, abnormally high >= 500 msec).
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: Double-blind safety analysis set (DB safety) included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 220 | 474
Participants
  Heart Rate value <=50 | 5 | 9
  Heart Rate value >=100 | 20 | 36
  PR Duration value >= 210 | 3 | 8
  QRS Duration value <= 50 | 0 | 0
  QRS Duration value >= 120 | 1 | 2
  QT Duration value <= 200 | 0 | 0
  QT Duration value >= 500 | 0 | 0

13. Secondary Outcome: Change From Baseline in the Body Mass Index (BMI) During DB Phase
Description: Change from baseline in BMI was reported.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 219 | 473
kilogram per meter square (kg/m^2) | 0.3 (1.78) | 0.0 (1.72)

14. Secondary Outcome: Change From Baseline in the Waist Circumference During DB Phase
Description: Change from baseline in waist circumference was reported.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 219 | 473
centimeter (cm) | 0.82 (5.137) | 0.37 (5.157)

15. Secondary Outcome: Change From Baseline in the Body Weight During DB Phase
Description: Change from baseline in body weight was reported.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 219 | 473
kilogram (kg) | 0.96 (5.103) | 0.10 (4.959)

16. Secondary Outcome: Change From Baseline in the Vital Signs (Pulse Rate) During DB Phase
Description: Change from baseline vital signs (pulse rate) were reported. This included supine pulse rate, standing pulse rate and supine-standing pulse rate.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Double-blind (DB) PP3M | Double-blind (DB) PP6M
Number analyzed (Participants) | 219 | 473
beats per minute (bpm)
  Supine Pulse Rate | 1.2 (11.57) | 0.6 (11.56)
  Standing Pulse Rate | 2.6 (12.28) | 0.9 (12.60)
  Pulse Rate (Standing-Supine) | 1.5 (8.85) | 0.2 (8.31)

17. Secondary Outcome: Change From Baseline in the Vital Signs (Systolic Blood Pressure [SBP] and Diastolic Blood Pressure [DBP]) During DB Phase
Description: Change from baseline in vital signs including SBP and DBP (supine/standing) were reported.
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Double-blind (DB) PP3M | Double-blind (DB) PP6M
Number analyzed (Participants) | 219 | 473
millimetre of mercury (mmHg)
  Supine SBP | -0.3 (13.14) | 0.6 (9.96)
  Standing SBP | 0.8 (12.08) | 1.3 (10.40)
  SBP (Standing-Supine) | 1.0 (9.83) | 0.6 (7.32)
  Supine DBP | 0.1 (9.25) | -0.4 (7.49)
  Standing DBP | 0.3 (9.39) | 0.4 (7.48)
  DBP (Standing-Supine) | 0.2 (7.79) | 0.7 (6.43)

18. Secondary Outcome: Change From Baseline in Positive and Syndrome Scale (PANSS) Subscales Score During DB Phase
Description: The neuropsychiatric symptoms of schizophrenia were assessed using the 30-item PANSS scale, which provides a total score (sum of the scores for all 30 items) and Scores for 3 subscales, that is, for positive subscale (sum of the scores of all 7 items) and negative subscale (sum of the scores of all 7 items) ranges from 7 (absent) to 49 (extreme psychopathology), and for the general psychopathology subscale (sum of the scores of all 16 items) score ranges from 16 (absent) to 112 (extreme psychopathology).
Time Frame: Baseline (DB) to 12 Months of DB Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 220 | 473
units on a scale
  Positive Subscale Score | -0.1 (2.82) | -0.1 (3.30)
  Negative Subscale Score | -0.6 (2.61) | -0.7 (2.70)
  General Psychopathology Subscale Score | -0.9 (4.18) | -1.0 (4.86)

19. Secondary Outcome: Number of Participants With Treatment-emergent Clinically Significant Abnormal Laboratory Values in Chemistry During DB Phase
Description: Number of participants with clinically significant abnormal laboratory values in chemistry included alanine aminotransferase (Unit per Litre [U/L]), albumin (Gram per Litre [g/L]), alkaline phosphatase (U/L), aspartate aminotransferase (U/L), bicarbonate (millimoles per litre [mmol/L]), bilirubin (micromoles per litre [umol/L]), calcium (mmol/L), chloride (mmol/L), cholesterol (mmol/L), creatinine (umol/L), gamma glutamyl transferase (GGT) (U/L), glucose (mmol/L), high-density lipoproteins (HDL) cholesterol (mmol/L), low density lipoproteins (LDL) cholesterol (mmol/L), lactate dehydrogenase (U/L), phosphate (mmol/L), potassium (mmol/L), protein (mmol/L), sodium (mmol/L), triglycerides (mmol/L), urate (umol/L), urea nitrogen (mmol/L) were reported. Here, ABL signifies abnormally low and ABH signifies abnormally high levels.
Time Frame: Up to 12 Months of DB Phase
Population: Double-Blind safety analysis set (DB safety) included all participants who were randomly assigned to treatment group of either PP6M or PP3M during the DB Phase and received at least 1 dose of PP6M/PP3M. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure. Here 'n' (number analyzed) included all evaluable participants who were analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 216 | 464
Participants
  Alanine Aminotransferase ABH | 0 | 1
  Albumin ABL | 0 | 0
  Albumin ABH | 0 | 0
  Alkaline Phosphatase ABH | 0 | 0
  Aspartate Aminotransferase ABH | 0 | 0
  Bicarbonate ABL | 0 | 3
  Bicarbonate ABH | 0 | 0
  Bilirubin ABH: number analyzed (Participants) | 208 | 447
  Bilirubin ABH | 0 | 1
  Calcium ABL | 0 | 0
  Calcium ABH | 0 | 0
  Chloride ABL: number analyzed (Participants) | 216 | 463
  Chloride ABL | 4 | 5
  Chloride ABH: number analyzed (Participants) | 216 | 463
  Chloride ABH | 0 | 0
  Cholesterol ABH: number analyzed (Participants) | 216 | 463
  Cholesterol ABH | 2 | 4
  Creatinine ABH | 0 | 0
  Gamma Glutamyl Transferase ABH | 0 | 2
  Glucose ABL | 1 | 0
  Glucose ABH | 1 | 5
  HDL Cholesterol ABL: number analyzed (Participants) | 216 | 463
  HDL Cholesterol ABL | 18 | 40
  LDL Cholesterol ABL: number analyzed (Participants) | 216 | 463
  LDL Cholesterol ABL | 33 | 44
  LDL Cholesterol ABH: number analyzed (Participants) | 216 | 463
  LDL Cholesterol ABH | 9 | 22
  Lactate Dehydrogenase ABH: number analyzed (Participants) | 215 | 456
  Lactate Dehydrogenase ABH | 0 | 1
  Phosphate ABL | 1 | 8
  Phosphate ABH | 0 | 0
  Potassium ABL: number analyzed (Participants) | 216 | 463
  Potassium ABL | 0 | 0
  Potassium ABH: number analyzed (Participants) | 216 | 463
  Potassium ABH | 0 | 0
  Protein ABL | 0 | 1
  Sodium ABL: number analyzed (Participants) | 216 | 463
  Sodium ABL | 1 | 0
  Sodium ABH: number analyzed (Participants) | 216 | 463
  Sodium ABH | 0 | 0
  Triglycerides ABH: number analyzed (Participants) | 216 | 463
  Triglycerides ABH | 4 | 6
  Urate ABL: number analyzed (Participants) | 215 | 463
  Urate ABL | 0 | 0
  Urate ABH: number analyzed (Participants) | 215 | 463
  Urate ABH | 1 | 4
  Urea Nitrogen ABH: number analyzed (Participants) | 215 | 464
  Urea Nitrogen ABH | 0 | 0

20. Secondary Outcome: Number of Participants With Treatment-emergent Clinically Significant Abnormal Laboratory Values in Hematology During DB Phase
Description: Number of participants with clinically significant abnormal laboratory values in hematology included hemoglobin (Hb), hematocrit (Hct), red blood cell (RBC) count, white blood cell (WBC) count with differential, platelets, hemoglobin A1c. Here, ABL signifies abnormally low and ABH signifies abnormally high levels.
Time Frame: Up to 12 Months of DB Phase
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | DB PP3M | DB PP6M
Number analyzed (Participants) | 215 | 459
Participants
  Basophils ABL | 0 | 0
  Eosinophils ABL | 1 | 1
  Erythrocytes ABL | 1 | 0
  Erythrocytes ABH | 0 | 0
  Hematocrit ABL: number analyzed (Participants) | 215 | 457
  Hematocrit ABL | 0 | 1
  Hematocrit ABH: number analyzed (Participants) | 215 | 457
  Hematocrit ABH | 0 | 0
  Hemoglobin ABL | 1 | 0
  Hemoglobin ABH | 0 | 0
  Leukocytes ABL | 0 | 0
  Leukocytes ABH | 2 | 4
  Lymphocytes ABL | 0 | 2
  Lymphocytes ABH | 1 | 1
  Monocytes ABH | 0 | 0
  Neutrophils ABL | 1 | 0
  Neutrophils ABH | 0 | 0
  Platelets ABL: number analyzed (Participants) | 214 | 458
  Platelets ABL | 0 | 0
  Platelets ABH: number analyzed (Participants) | 214 | 458
  Platelets ABH | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2.5 Years
Description: Open-label (OL) safety set included all participants who received at least 1 dose of OL study drug (excluding the first study participants if re-screened), both transition and maintenance phases. Double-blind (DB) safety set included all participants who were randomly assigned to treatment group either PP6M or PP3M during DB Phase and received at least 1 dose of DB study drug. Participants from DB safety set continued in follow-up phase.
Arm/Group | Open-Label (OL) PP1M/PP3M | Double-blind PP3M | Double-blind PP6M | Follow-up (FU) Phase PP3M | Follow-up Phase PP6M
All-Cause Mortality (participants affected / at risk) | 1/838 | 2/224 | 1/478 | 0/42 | 0/109
Serious Adverse Events (participants affected / at risk) | 23/838 | 15/224 | 24/478 | 1/42 | 6/109
Other Adverse Events (participants affected / at risk) | 127/838 | 52/224 | 125/478 | 1/42 | 5/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label (OL) PP1M/PP3M (N=838) | Double-blind PP3M (N=224) | Double-blind PP6M (N=478) | Follow-up (FU) Phase PP3M (N=42) | Follow-up Phase PP6M (N=109)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden Death (General disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Nasal Sinus Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Acute Psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Adjustment Disorder with Mixed Anxiety and Depressed Mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Adjustment Disorder with Mixed Disturbance of Emotion and Conduct (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Behavioural Addiction (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination, Auditory (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mixed Anxiety and Depressive Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Panic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 3 | 2 | 1 | 0 | 0
Psychotic Symptom (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 6 | 1 | 8 | 0 | 2
Suicidal Ideation (Psychiatric disorders) | 3 | 2 | 1 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 2 | 0 | 2 | 0 | 1
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Mammoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Artery Occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label (OL) PP1M/PP3M (N=838) | Double-blind PP3M (N=224) | Double-blind PP6M (N=478) | Follow-up (FU) Phase PP3M (N=42) | Follow-up Phase PP6M (N=109)
Injection Site Pain (General disorders) | 72 | 9 | 37 | 0 | 0
Nasopharyngitis (Infections and infestations) | 22 | 13 | 22 | 1 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 9 | 24 | 0 | 1
Weight Increased (Investigations) | 8 | 17 | 40 | 0 | 0
Headache (Nervous system disorders) | 16 | 12 | 32 | 0 | 0

LIMITATIONS AND CAVEATS:
The non-inferiority design was based on the principle of enrichment; that is, criteria of clinical stability were applied prior to entry into the Double-blind Phase. Hence, the ITT (DB) analysis set does not reflect the overall sample of participants who were initially enrolled in Study PSY3015 (ClinicalTrials.gov Identifier: NCT03345342) for treatment with PP3M/PP6M. Therefore, results may not reflect true efficacy for prevention of relapses in the overall population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the Sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT03345342/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03345342/SAP_001.pdf